CLINICAL TRIAL: NCT01838174
Title: A Phase IV Trial of Neuroprotection With ACTH in Acute Optic Neuritis
Brief Title: A Trial of Neuroprotection With ACTH in Acute Optic Neuritis
Acronym: ACTHAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor requested
Sponsor: University of Colorado, Denver (Other)
Collaborators: Mallinckrodt (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0388
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis
Keywords: Optic Neuritis
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis | interventions — Adrenocorticotropic Hormone; Methylprednisolone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acthar Gel (ACTH) (Experimental): 15 days of intramuscular (IM) or sub-cutaneous corticotropin (SQ) Acthar (ACTH).
  Interventions: Drug: ACTHAR Gel (ACTH)
- IV methylprednisolone (steroids) (Active Comparator): 3 days of IV methylprednisolone (steroids) followed by 11 days of oral prednisone
  Interventions: Drug: IV methylprednisolone (steroids)

INTERVENTIONS:
Drug: ACTHAR Gel (ACTH) — 15 days of daily injections
  Other Names: ACTH
  Arms: Acthar Gel (ACTH)
Drug: IV methylprednisolone (steroids) — 3 days of intravenous methylprednisolone followed by 11 days of oral taper
  Other Names: methylprednisolone
  Arms: IV methylprednisolone (steroids)

SUMMARY:
We hypothesize that the novel melanocortin-mediated anti-inflammatory effects of ACTH will reduce axonal loss following ON by limiting inflammatory optic nerve injury. We will compare the effect of ACTH and intravenous methylprednisolone therapy on axonal injury following ON using OCT, a sensitive, reproducible and noninvasive tool to measure RNFL thickness.

The primary outcome will be the average RNFL thickness at 6 months. Additional pre-specified statistical analyses will compare the difference in the mean RNFL thickness at 6 months in the affected eye between the IV methylprednisolone- and Acthar-treated groups, and the mean 6-month affected eye RNFL thicknesses adjusted for the baseline unaffected eye RNFL. The secondary outcome measure will examine the frequency of optic nerves with RNFL swelling between the IV methylprednisolone- and Acthar-treated groups at 1 and 3 months. A predefined exploratory outcome will compare the ganglion cell plus inner plexiform layer (GC+IPL) thickness at 6 months between treatment groups. Additional tertiary outcome will be the assessment of changes in fatigue, mood, visual function depression, and quality of life in patients with AON. Assessment will be completed by administration of the following questionnaires: Modified Fatigue Impact Scale, Multiple Sclerosis Quality of Life 54 Instrument, 25-item Visual Function Questionnaire with 10-item supplement, Beck's Depression Inventory. These questionnaires have been validated for the MS (AON) population. Descriptive and correlative analysis will be done at each visit time point to assess for QOL for this study population.

DETAILED DESCRIPTION:
Patients with their first episode of unilateral acute ON will be treated with either 3 days of IV methylprednisolone followed by 11 days of oral prednisone or 15 days of intramuscular or subcutaneous corticotropin (Acthar).

This is a parallel active group, randomized controlled trial in which up to 100 people with clinically unilateral acute optic neuritis (≤ 2 weeks of vision loss; with or without a previous diagnosis of relapsing remitting MS) will be treated with either ACTH or IV methylprednisolone/prednisone for 2 weeks to assess RNFL thickness. The primary, secondary, and tertiary outcomes will be as noted above. Participants will be assessed for inclusion/exclusion criteria by their treating neurologist/ophthalmologist at the University of Colorado Denver (PI- Dr. Jeffrey Bennett) or The University of Pennsylvania Scheie Eye Institute (PI- Dr. Kenneth Shindler). Following informed consent, the University of Colorado will determine patient randomization for both sites per the established randomization scheme. A secured fax or email confirmation regarding randomization will be sent to the University of Pennsylvania research staff and proper pharmacy orders will be placed by the site investigator or designee. We expect to enroll up to 50 subjects per institution.

Following informed consent and randomization, participants will undergo baseline procedures (visit 1) and receive treatment with either high dose methylprednisolone (1000 mg IV qD for 3 days followed by 60 mg oral prednisone daily for 11 days) or Acthar (80 U IM or SC daily for 5 days followed by 40 U IM or SC daily for 10 days). Study follow-up visits will subsequently occur at 1, 3, and 6 months. During each visit, including baseline (visit 1), ETDRS, low contrast acuity (2.5%), and color vision (Farnsworth D-15) will be assessed. OCT evaluations (Optic Disc Cube 200x200 and Macular Cube 512x128) will be performed at baseline, 1, 3 and 6 months using spectral domain OCT (Cirrus OCT; Carl Zeiss Meditec, Dublin, CA, USA). Automated visual fields (Humphrey 30-2 SITA) will be performed at baseline (visit 1) and month 6. Modified Fatigue Impact Scale, Multiple Sclerosis Quality of Life 54 Instrument, 25-item Visual Function Questionnaire with 10-item supplement, Beck's Depression Inventory questionnaires will be assessed at each study visit. The patient's treating physician will perform blood tests and MRI evaluations to exclude other causes of optic neuropathy at the initial study visit as part of their routine care.

RNFL edema will be defined as either average RNFL thickness greater than the 95th percentile of the age matched normal database or a ratio of RNFL thickness (affected/fellow eye) greater than 1.1 in any quadrant.8 The study sites will collect and report data on AEs and SAEs per standard practice.

Detailed Patient Schedule of Assessments:

Baseline, within 2 weeks of onset of vision loss (approximately 2 hours):

* Consent and Discussion of Study Expectations
* Eligibility Checklist
* Review of Medical History & Demographics
* Record list of Con Meds, Co-Morbidities, and Symptoms at time of Diagnosis
* Obtain Randomization Number
* Administer MFIS, BDI, VFQ-25 and 10-item supplement, and MSQOL-54 questionnaires
* Eye Testing (OCT - [Optic Disc Cube 200x200 and Macular Cube 512x128], Visual Acuity [High Contrast ETDRS], Low-contrast Letter Acuity [Sloan 2.5% and 1.25% letters], Color Vision [Farnsworth D15], Humphrey's visual fields (HVF).
* Administer Study Medication (either IM or SC Acthar Gel or IV Methylprednisolone with oral taper)
* Labs and MRI, per standard of care

Month 1 +/- 3 days (approximately 1.5 hours):

* Review of AEs and Con Meds
* Administer MFIS, BDI, VFQ-25 and 10-item supplement, and MSQOL-54 questionnaires
* Eye Testing (OCT - [Optic Disc Cube 200x200 and Macular Cube 512x128], Visual Acuity [High Contrast ETDRS], Low-contrast Letter Acuity [Sloan 2.5% and 1.25% letters], Color Vision [Farnsworth D15]

Month 3 +/- 3 days (approximately 1.5 hours):

* Review of AEs and Con Meds
* Administer MFIS, BDI, VFQ-25 and 10-item supplement, and MSQOL-54 questionnaires
* Eye Testing (OCT - [Optic Disc Cube 200x200 and Macular Cube 512x128], Visual Acuity [High Contrast ETDRS], Low-contrast Letter Acuity [Sloan 2.5% and 1.25% letters], Color Vision [Farnsworth D15]

Month 6 +/- 3 days (approximately 2 hours):

* Review of AEs and Con Meds
* Administer MFIS, BDI, VFQ-25 and 10-item supplement, and MSQOL-54 questionnaires
* Eye Testing (OCT - [Optic Disc Cube 200x200 and Macular Cube 512x128], Visual Acuity [High Contrast ETDRS], Low-contrast Letter Acuity [Sloan 2.5% and 1.25% letters], Color Vision [Farnsworth D15], Humphrey's visual fields (HVF)

ELIGIBILITY:
Inclusion criteria

1. Ability to provide written informed consent before any study assessment is performed.
2. Male and female patients aged between 18 and 55 years, inclusive.
3. Diagnosis of clinically unilateral acute demyelinating optic neuritis (ADON)
4. Clinical signs and symptoms of ADON starting within the 14 day prior to intended randomization (loss of vision, pain on movement, impairment of color vision).
5. The qualifying episode of optic neuritis must be the first clinical episode of optic neuritis in the affected eye.
6. Able to undergo treatment with intravenous methylprednisolone or Acthar gel.

Exclusion Criteria:

1. Functionally or clinically relevant comorbidity of the affected eye (e.g., glaucoma, amblyopia, optic nerve hypoplasia, macular hole, macular edema, vitreomacular traction, uveitis, diabetes, optic neuritis, or other diseases of the optic nerve or a history thereof).
2. Bilateral optic neuritis.
3. Concurrent functionally or clinically relevant disturbances of the eye not affected by ADON.
4. High clinical likelihood of a form of optic neuritis other than ADON (e.g., no pain on movement, no light perception, severe optic disk edema, atrophic optic disk, retinal exudates, or hemorrhages).
5. Non-assessable OCT at screening.
6. Refractive error greater than ±5 diopters or (pre-surgical value to be used for patients having undergone refractive surgery).
7. Patients with an immune system disorder other than MS or ADON (e.g. rheumatoid arthritis, scleroderma, Sjogren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with a known immunodeficiency syndrome (AIDS, hereditary immune deficiency, drug-induced immune deficiency). Diagnosis of neuromyelitis optica or MOG-IgG will not exclude a patient from the study but will be accounted for in the data analysis.
8. Prior treatment with IVMP or Acthar gel within the past 30 days.
9. Treatment with, mitoxantrone, cyclophosphamide, mycophenolate, azathioprine, or other non-approved agents for the treatment of relapsing forms of MS.
10. Concurrent use of 4-aminopyridine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05; Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Retinal Nerve Fiber Layer (RNFL) thickness | 6 months
  The primary outcome will be the average RNFL thickness at 6 months.

SECONDARY OUTCOMES:
Frequency of RNFL swelling | 1 and 3 months
  The secondary outcome measure will examine the frequency of optic nerves with RNFL swelling between the IV methylprednisolone- and Acthar-treated groups at 1 and 3 months.

OTHER OUTCOMES:
Comparison of ganglion cell plus inner plexiform layer (GC+IPL) thickness at 6 months | 6 months
  Exploratory outcome will compare the ganglion cell plus inner plexiform layer (GC+IPL) thickness at 6 months between treatment groups
Assessment of changes in fatigue in patients with AON. | Baseline, Month 1, 3, 6
  Assessment will be completed by administration of the following questionnaire: Modified Fatigue Impact Scale. This questionnaire has been validated for the MS (AON) population. Descriptive and correlative analysis will be done at each visit time point to assess for QOL for this study population.
Assessment in mood in patients with AON. | Baseline, Month 1, 3, 6
  Assessment will be completed by administration of the following questionnaire: Multiple Sclerosis Quality of Life 54 Instrument. This questionnaire has been validated for the MS (AON) population. Descriptive and correlative analysis will be done at each visit time point to assess for QOL for this study population.
Assessment in visual function in patients with AON. | Baseline, Month 1, 3, 6
  Assessment will be completed by administration of the following questionnaires: 25-item Visual Function Questionnaire with 10-item supplement.
Assessment in quality of life in patients in patients with AON. | Baseline, Month 1, 3, 6
  Assessment will be completed by administration of the following questionnaire: Beck's Depression Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bennett, MD, PhD, Principal Investigator — University of Colorado, Denver; Kenneth Shindler, MD, PhD, Principal Investigator — University of Pennsylvania Scheie Eye Institute
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennett JL, Grove NC, Johnson RK, Mizenko C, DuPont JC, Wagner BD, Lynch AM, Frohman TC, Shindler KS, Frohman EM. A Randomized Prospective Trial Comparing Repository Corticotropin Injection and Intravenous Methylprednisolone for Neuroprotection in Acute Optic Neuritis. J Neuroophthalmol. 2023 Sep 1;43(3):323-329. doi: 10.1097/WNO.0000000000001878. Epub 2023 Jun 1. PMID 37261907